CLINICAL TRIAL: NCT05827523
Title: Phase III Randomized Trial of HIPEC in Primary Stage Three & Four Primary Ovarian Cancer After Interval Cytoreductive Surgery (FOCUS, KOV-04)
Brief Title: Interval Cytoreductive Surgery With or Without HIPEC for Ovarian Cancer
Acronym: FOCUS / KOV-04
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Myong Cheol Lim, MD, PhD, Principal Researcher, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCC2023-0100
Record Dates: First submitted 2023-04-12; First posted 2023-04-25 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Ovarian Cancer
Keywords: Ovarian cancer; Hyperthermic intraperitoneal chemotherapy; HIPEC; Interval cytoreductive surgery; Neoadjuvant chemotherapy; Carcinoma, Ovarian Epithelial; Epithelial ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Cisplatin

STUDY DESIGN:
Intervention Model Description: Randomized controlled, single-blinded, multicenter phase III trial
Who Masked: Participant
Masking Description: Enrolled patients are unaware of which group they have been assigned to.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- HIPEC (Experimental): Interval cytoreductive surgery with HIPEC
  Interventions: Drug: Cisplatin
- No HIPEC (No Intervention): Interval cytoreductive surgery without HIPEC

INTERVENTIONS:
Drug: Cisplatin — Hyperthermic intraperitoneal chemotherapy (HIPEC) with cisplatin 75mg/m2 after interval cytoreductive surgery
  Arms: HIPEC

SUMMARY:
Primary stage III-IV epithelial ovarian cancer randomizing between interval cytoreductive surgery with or without hyperthermic intraperitoneal chemotherapy (HIPEC)

DETAILED DESCRIPTION:
The goal of this phase III randomized controlled trial is to compare the clinical efficacy of HIPEC with cisplatin (trial arm) compared to no HIPEC (control arm) during interval cytoreductive surgery followed by neoadjuvant chemotherapy, in patients with stage III-IV primary epithelial ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and written informed consent,
2. Patients ≥18, <80 years old,
3. Diagnosed with histologically confirmed FIGO stage III-IV primary epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer treated with three cycles of neoadjuvant chemotherapy,
4. Treated with interval complete cytoreduction, or cytoreduction with no more than 2.5 mm depth of residual disease,
5. A life expectancy > 3 months as clinically judged,
6. Adequate organ function for cytoreductive surgery and HIPEC,
7. Women who are medically unable to conceive or who are of childbearing potential, agree to follow contraceptive guidelines during treatment and,
8. Patients can also consent to the provision of clinical information for secondary use, such as future biomedical research. However, in the future, subjects can participate in the main trial even if they do not intend to participate in sharing clinical information.

Exclusion Criteria:

1. Diagnosed with non-epithelial ovarian carcinoma or borderline ovarian tumor
2. Patients who have not undergone neoadjuvant chemotherapy,
3. Interval cytoreduction with more than 2.5 mm depth of residual disease,
4. A life expectancy ≤3 months as clinically judged,
5. History of previous malignancy within five years prior to inclusion, that affects ovarian cancer treatment results, with the exception of carcinoma in situ, radically excised basal cell or squamous cell cancer of the skin, or synchronal endometrial carcinoma FIGO IA G1/2,
6. Patients with myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or with features suggestive of MDS/AML,
7. Patients with active central nervous system metastasis and carcinoma meningitis or patients who have been previously treated for brain metastases must be in a stable state in radiology,
8. Patients with antibacterial, antifungal, or antiviral infections requiring systemic treatment (administration of parenteral antibiotics),
9. Active tuberculosis that is not controlled within 1 month of treatment,
10. Patients diagnosed with a psychiatric disorder or substance abuse disorder that would interfere with your ability to cooperate with the trial,
11. Patients with any contraindications to the use of cisplatin (i.e., hypersensitivity to cisplatin),
12. Patients with a history of allogeneic tissue/solid organ transplantation or bone marrow transplantation or a history of double umbilical cord transplantation or,
13. History or current evidence of any condition, therapy, or laboratory abnormality that may confound the results of the study, or interfere with the patient's participation, in the opinion of the treating investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From randomization to the date of death from any cause, assessed up to 5 years

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From randomization to time of first progression or death from any cause, whichever came first, assessed up to 5 years
Cancer-specific survival | From randomization to the date of death due to ovarian cancer, assessed up to 5 years
Time to first subsequent therapy (TFST) | from the last day of the last cycle of a prior regimen of chemotherapy to the first day of the first cycle of the subsequent chemotherapy, assessed up to 5 years
  the interval from the last day of the last cycle of a prior regimen of chemotherapy to the first day of the first cycle of the subsequent regimen for each course of chemotherapy
Treatment-related adverse events | From randomization up to the end of treatment plus 4 weeks
  assessed by CTCAE ver.5.0
Health-related quality of life (EORTC-QLQ-C30) | Over the 5 year surveillance period
  The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to the questions are scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better overall health status.
Health-related quality of life (EORTC-QLQ-OV28) | Over the 5 year surveillance period
  The EORTC QLQ-OV28 is a specified questionnaire for patients with ovarian cancer. Participant responses to the question are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized so that scores range from 0 to 100. A lower score indicates a better outcome.
Health-related quality of life (EQ-5D-5L) | Over the 5 year surveillance period
  Each dimension in the EQ-5D-5L has five response levels: no problems (Level 1); slight; moderate; severe; and extreme problems (Level 5).
Cost-effectiveness analysis | At time of completion of 5-year surveillance period
  assessed by Quality-Adjusted Live Years (QALYs), incremental cost-effectiveness ratio (ICER)

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No